CLINICAL TRIAL: NCT00137358
Title: Phase I Trial of Dose Escalated IMRT to the Para-aortic Nodes With Concurrent Cisplatin and Amifostine in Locally Advanced Cervical Cancer
Brief Title: Radiation With Chemotherapy and a Study Drug to the Para-Aortic Nodes in Cervical Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: unable to obtain funding to conduct study
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Principal Investigator, Jennifer F. De Los Santos, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETH175-04D
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Cervical Cancer
Keywords: Cervical; Uterine; Para-aortic; Nodes; IMRT; Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms | interventions — Radiotherapy; Cisplatin; Amifostine

INTERVENTIONS:
Procedure: Radiation Therapy
Drug: Cisplatin
Drug: Amifostine

SUMMARY:
Investigator has since decided not to pursue this protocol further. No patients were enrolled.

This study is to determine the maximum tolerated dose of external beam radiation to the para-aortic lymph nodes using intensity modulated radiation therapy (IMRT).

This protocol will test the hypothesis that the use of IMRT and amifostine will decrease GI toxicity and therefore allow the radiation dose to the para-aortic lymph nodes to be safely escalated.

DETAILED DESCRIPTION:
This is a Phase I open-label multi-institutional study that will enroll a minimum of 27 and up to 42 patients with locally advanced cervical cancer (a minimum of 27 will be entered if all dose levels are explored without reaching a dose limiting toxicity at any level). The primary objective is to determine the maximum tolerated dose (MTD) of external beam radiation to the para-aortic lymph nodes using IMRT and amifostine. Patients will be stratified according to gross tumor volume (GTV) prior to dose escalation.

Within each GTV stratum, the dose escalation will be determined as follows: Accrue 3 patients in the first dose level based on the determined stratum. A Dose Limiting Toxicity is defined as the development of > Grade 3 acute GI toxicity, per the RTOG acute toxicity scale. If no DLT is observed at the first dose level, 3 patients will be enrolled at the next dose level. If one patient experiences DLT at a given dose level, 3 additional patients will be enrolled at that dose level. If 0 of these 3 additional patients experience DLT, dosing of the next dose level is begun. If 1 or more of these 3 additional patients experience DLT at the highest dose level below the maximally administered dose, this dose becomes the recommended dose. At least 6 patients must be entered at this recommended dose. The Maximum Tolerated Dose (MTD) is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* No prior therapy other than biopsy of the cervix or endoscopic pelvic nodal resection.
* Patients may have endoscopic resection of enlarged pelvic and low common iliac nodes, however, needle biopsy only of enlarged para-aortic nodes will be eligible for entry.
* Patients with squamous cell, adenocarcinoma, and adenosquamous carcinoma are eligible.
* Patients must have no evidence of metastatic disease outside of the pelvis (except to the para-aortic nodes).
* Patients must have Zubrod performance status 0-1 and no medical contraindications to the administration of full dose chemotherapy.
* Patients must have a life expectancy > 6 months
* Adequate bone marrow function: white blood cell (WBC) 3000/mm3 (absolute neutrophil count [ANC] 1500/mm3); adequate renal function: creatinine 1.5 mg/dl (urinary diversion is permitted to improve renal function); patients must have bilirubin 1.5 mg/dl, ALT 2 x normal.
* No prior (within last 3 years) or simultaneous malignancies (other than basal cell or non-invasive tumors)

Exclusion Criteria:

* Complete resection of the involved para-aortic nodes.
* Patients with evidence of bowel adherent to the GTV by contrast enhanced computed tomography (CT) scan will be ineligible.
* Patients with the following histologies will be ineligible: glassy cell, small cell, carcinoid, adenoid cystic, and clear cell.
* Prior (within last 3 years) malignancies other than basal cell carcinoma or non-invasive malignancies.
* Prior chemotherapy.
* Prior pelvic or abdominal radiation (other than transvaginal irradiation to control bleeding).
* Prior tumor-directed surgery other than lymph node sampling/staging
* Life expectancy < 6 months
* Patients who are pregnant will be ineligible.
* Patients with insulin dependent diabetes will be ineligible.
* Patients who are obese, such that reliable immobilization is not achieved.
* Patients with pain or discomfort that would preclude lying still for extended periods of time.
* Patients with tumors that are bleeding and require more immediate treatment.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the maximum tolerated dose (MTD) of external beam radiation to the para-aortic lymph nodes using IMRT and amifostine.

SECONDARY OUTCOMES:
The secondary endpoints include local-regional control, overall survival and toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer F De Los Santos, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Grigsby PW, Heydon K, Mutch DG, Kim RY, Eifel P. Long-term follow-up of RTOG 92-10: cervical cancer with positive para-aortic lymph nodes. Int J Radiat Oncol Biol Phys. 2001 Nov 15;51(4):982-7. doi: 10.1016/s0360-3016(01)01723-0. PMID 11704321
- [Background] Berman ML, Keys H, Creasman W, DiSaia P, Bundy B, Blessing J. Survival and patterns of recurrence in cervical cancer metastatic to periaortic lymph nodes (a Gynecologic Oncology Group study). Gynecol Oncol. 1984 Sep;19(1):8-16. doi: 10.1016/0090-8258(84)90151-3. PMID 6469092
- [Background] Lepanto P, Littman P, Mikuta J, Davis L, Celebre J. Treatment of para-aortic nodes in carcinoma of the cervix. Cancer. 1975 Jun;35(6):1510-3. doi: 10.1002/1097-0142(197506)35:63.0.co;2-u. PMID 807311
- [Background] Lovecchio JL, Averette HE, Donato D, Bell J. 5-year survival of patients with periaortic nodal metastases in clinical stage IB and IIA cervical carcinoma. Gynecol Oncol. 1989 Jul;34(1):43-5. doi: 10.1016/0090-8258(89)90103-0. PMID 2737524
- [Background] Nori D, Valentine E, Hilaris BS. The role of paraaortic node irradiation in the treatment of cancer of the cervix. Int J Radiat Oncol Biol Phys. 1985 Aug;11(8):1469-73. doi: 10.1016/0360-3016(85)90334-7. PMID 4019270
- [Background] Tewfik HH, Buchsbaum HJ, Latourette HB, Lifshitz SG, Tewfik FA. Para-aortic lymph node irradiation in carcinoma of the cervix after exploratory laparotomy and biopsy-proven positive aortic nodes. Int J Radiat Oncol Biol Phys. 1982 Jan;8(1):13-8. doi: 10.1016/0360-3016(82)90378-9. PMID 7061247
- [Background] Grigsby PW, Perez CA, Chao KS, Herzog T, Mutch DG, Rader J. Radiation therapy for carcinoma of the cervix with biopsy-proven positive para-aortic lymph nodes. Int J Radiat Oncol Biol Phys. 2001 Mar 1;49(3):733-8. doi: 10.1016/s0360-3016(00)00806-3. PMID 11172956
- [Background] Rubin SC, Brookland R, Mikuta JJ, Mangan C, Sutton G, Danoff B. Para-aortic nodal metastases in early cervical carcinoma: long-term survival following extended-field radiotherapy. Gynecol Oncol. 1984 Jun;18(2):213-7. doi: 10.1016/0090-8258(84)90028-3. PMID 6735264
- [Background] Carl UM, Bahnsen J, Wiegel T. Radiation therapy of para-aortic lymph nodes in cancer of the uterine cervix. Acta Oncol. 1993;32(1):63-7. doi: 10.3109/02841869309083887. PMID 8466766
- [Background] Varia MA, Bundy BN, Deppe G, Mannel R, Averette HE, Rose PG, Connelly P. Cervical carcinoma metastatic to para-aortic nodes: extended field radiation therapy with concomitant 5-fluorouracil and cisplatin chemotherapy: a Gynecologic Oncology Group study. Int J Radiat Oncol Biol Phys. 1998 Dec 1;42(5):1015-23. doi: 10.1016/s0360-3016(98)00267-3. PMID 9869224
- [Background] Podczaski E, Stryker JA, Kaminski P, Ndubisi B, Larson J, DeGeest K, Sorosky J, Mortel R. Extended-field radiation therapy for carcinoma of the cervix. Cancer. 1990 Jul 15;66(2):251-8. doi: 10.1002/1097-0142(19900715)66:23.0.co;2-e. PMID 2369710
- [Background] Malfetano JH, Keys H. Aggressive multimodality treatment for cervical cancer with paraaortic lymph node metastases. Gynecol Oncol. 1991 Jul;42(1):44-7. doi: 10.1016/0090-8258(91)90228-w. PMID 1916509
- [Background] Mutic S, Malyapa RS, Grigsby PW, Dehdashti F, Miller TR, Zoberi I, Bosch WR, Esthappan J, Low DA. PET-guided IMRT for cervical carcinoma with positive para-aortic lymph nodes-a dose-escalation treatment planning study. Int J Radiat Oncol Biol Phys. 2003 Jan 1;55(1):28-35. doi: 10.1016/s0360-3016(02)03804-x. PMID 12504033
- [Background] Aoki T, Nagata Y, Mizowaki T, Kokubo M, Negoro Y, Takayama K, Mitsumori M, Sasai K, Hiraoka M. Clinical evaluation of dynamic arc conformal radiotherapy for paraaortic lymph node metastasis. Radiother Oncol. 2003 Apr;67(1):113-8. doi: 10.1016/s0167-8140(02)00388-2. PMID 12758247
- [Background] Wadler S, Goldberg G, Fields A, Anderson P, Beitler JJ, Sood B, Haynes H, Runowicz C. The potential role of amifostine in conjunction with cisplatin in the treatment of locally advanced carcinoma of the cervix. Semin Oncol. 1996 Aug;23(4 Suppl 8):64-8. PMID 8783670
- [Background] Gallardo D, Mohar A, Calderillo G, Mota A, Solorza G, Lozano A, Solano P, De La Garza J. Cisplatin, radiation, and amifostine in carcinoma of the uterine cervix. Int J Gynecol Cancer. 1999 May;9(3):225-230. doi: 10.1046/j.1525-1438.1999.99029.x. PMID 11240771
- [Background] Koukourakis MI, Kyrias G, Kakolyris S, Kouroussis C, Frangiadaki C, Giatromanolaki A, Retalis G, Georgoulias V. Subcutaneous administration of amifostine during fractionated radiotherapy: a randomized phase II study. J Clin Oncol. 2000 Jun;18(11):2226-33. doi: 10.1200/JCO.2000.18.11.2226. PMID 10829042
- [Background] Athanassiou H, Antonadou D, Coliarakis N, Kouveli A, Synodinou M, Paraskevaidis M, Sarris G, Georgakopoulos GR, Panousaki K, Karageorgis P, Throuvalas N; Oncology Hellenic Group. Protective effect of amifostine during fractionated radiotherapy in patients with pelvic carcinomas: results of a randomized trial. Int J Radiat Oncol Biol Phys. 2003 Jul 15;56(4):1154-60. doi: 10.1016/s0360-3016(03)00187-1. PMID 12829154